CLINICAL TRIAL: NCT02840097
Title: Traumatic Injury Clinical Trial Evaluating Tranexamic Acid in Children (TIC-TOC): A Pilot and Feasibility Study
Brief Title: Traumatic Injury Clinical Trial Evaluating Tranexamic Acid in Children: A Pilot and Feasibility Study
Acronym: TIC-TOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daniel Nishijima, MD, MAS (Other)
Collaborators: Pediatric Emergency Care Applied Research Network (Network)
Responsible Party: Sponsor-Investigator, Daniel Nishijima, MD, MAS, Associate Professor, Emergency Medicine, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1023599
Record Dates: First submitted 2016-07-14; First posted 2016-07-21 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Brain Injuries; Wounds and Injuries; Hemorrhage
Keywords: Brain injuries; Wounds and injuries; Hemorrhage; Tranexamic acid; Child
MeSH Terms: conditions — Brain Injuries; Wounds and Injuries; Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tranexamic acid dose A (Experimental): Subjects will receive a 15 mg/kg bolus of tranexamic acid over 10 minutes followed by a 2mg/kg/h over 8 hours. This represents 31mg/kg total dose of TXA.
  Interventions: Drug: Tranexamic Acid
- Tranexamic acid dose B (Experimental): Subjects will receive a 30 mg/kg bolus of tranexamic acid over 10 minutes followed by a 4 mg/kg/h over 8 hours. This represents 62 mg/kg total dose of TXA.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Subjects in the placebo group will receive a bolus dose of normal saline over 10 minutes followed by a normal saline infusion over 8 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Active drug is provided to participants as described based on the TXA arm they are randomized to.
  Other Names: TXA
  Arms: Tranexamic acid dose A; Tranexamic acid dose B
Drug: Placebo — Normal saline is provided to participants if randomized to this treatment arm.
  Other Names: 0.9% Normal Saline
  Arms: Placebo

SUMMARY:
Trauma is the leading cause of death and disability in children in the United States. The long-term goal of this project is to evaluate the benefits and harms of tranexamic acid (TXA; a drug that stops bleeding) in severely injured children. This is a 40-patient pilot study to evaluate the feasibility of two subsequent large-scale studies of TXA in injured children.

DETAILED DESCRIPTION:
Tranexamic acid (TXA), a drug that stops bleeding, is the only drug treatment that improves survival in adults with serious bleeding after injuries. However, TXA has not been used routinely in children with traumatic bleeding because no studies have appropriately evaluated TXA for injured children. Such a study has the potential for significant impact in improving the lives of injured children and their families, if found to be successful. The long-term objective is to evaluate the benefits and risks of TXA in severely injured children. This will be achieved by ultimately conducting two large-scale, multicenter, randomized controlled trials of TXA use in severely injured children. One trial will evaluate TXA in children with severe injuries to the body ("torso injuries", i.e., to the abdomen and chest) and the second trial will evaluate TXA in children with moderate-to-severe traumatic brain injuries (TBIs). However, conducting a clinical trial in critically ill children is challenging due to lower disease frequency and complex parent consent/child assent procedures. The investigators will conduct a pilot study, designed similarly to the full-scale trials but with much smaller patient enrollment, to assess the feasibility of, and fill crucial information gaps for the two subsequent large-scale clinical trials. Injured children will be randomized to one of three study arms: two different TXA doses or placebo. The specific aim of the proposed pilot study is to demonstrate the ability to efficiently identify and enroll children with hemorrhagic torso injuries or TBIs into a multicenter, randomized controlled pilot study evaluating these two doses of TXA and placebo. The pilot study will enroll 40 children who meet inclusion and exclusion criteria at 4 participating sites. To demonstrate the ability to collect outcome measures, the investigators will collect the identical anticipated outcome measures for the subsequent clinical trials: total blood products transfused over the initial 48 hours of care (torso injury trial), and intracranial hemorrhage progression in first 24 hours and neurocognitive function at 6 months after randomization (TBI trial). The investigators will also collect safety outcomes, specifically venothromboembolic events (i.e., blot clots in the blood vessels) and seizures within the initial 24 hours of study drug. Additional objectives of this pilot study are to: evaluate the ability to efficiently screen, identify, consent, randomize, and initiate the study intervention within 3 hours of injury, assess protocol adherence and variability of care in enrolled patients, and identify operational efficiencies with the potential to enhance the success of the subsequent trials.

ELIGIBILITY:
Inclusion Criteria:

1. Less than 18 years old AND
2. Penetrating torso trauma, blunt torso trauma, or head trauma as defined below.
3. Penetrating Torso Trauma:

   a. Penetrating trauma to the chest, abdomen, neck, pelvis or thigh with at least one of the following:
   * age-adjusted hypotension, or
   * age-adjusted tachycardia despite adequate resuscitation fluids, or
   * radiographic evidence of internal hemorrhage, or
   * clinician suspicion of ongoing internal hemorrhage
4. Blunt Torso Trauma (at least one of the following):

   1. Clinician suspicion of hemorrhagic blunt torso injury and at least one of the following:

      * age-adjusted hypotension, or
      * persistent age-adjusted tachycardia despite adequate resuscitation fluids
   2. Hemothorax on chest tube placement or imaging,
   3. Clinical suspicion of hemorrhagic blunt torso injury and Intraperitoneal fluid on abdominal ultrasonography (Focused Assessment with Sonography in Trauma),
   4. Intra-abdominal injury on CT with either contrast extravasation or more than trace intraperitoneal fluid,
   5. Pelvic fracture with contrast extravasation or hematoma on abdominal/pelvic CT scan with at least one of the following:

      * Age-adjusted tachycardia, or
      * Age-adjusted hypotension.
5. Head Trauma:

   1. Initial Glasgow Coma Scale (GCS) score 3 to 13 with associated intracranial hemorrhage on cranial CT scan (enroll after cranial CT scan)

Exclusion Criteria:

1. Unable to administer study drug within 3 hours of traumatic event
2. Known pregnancy
3. Known prisoners
4. Known wards of the state
5. Cardiac arrest prior to randomization
6. GCS score of 3 with bilateral unresponsive pupils
7. Isolated subarachnoid hemorrhage, epidural hematoma, or diffuse axonal injury
8. Known bleeding/clotting disorders
9. Known seizure disorders
10. Known history of severe renal impairment
11. Unknown time of injury
12. Previous enrollment into the TIC-TOC trial
13. Prior TXA for current injury
14. Non-English and non-Spanish speaking
15. Known venous or arterial thrombosis

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2020-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K Nishijima, MD, MAS, Principal Investigator — University of California, Davis
Locations (4):
- United States (4):
  - University of California, Davis, Sacramento, California
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nishijima DK, VanBuren J, Hewes HA, Myers SR, Stanley RM, Adelson PD, Barnhard SE, Bobinski M, Ghetti S, Holmes JF, Roberts I, Schalick WO 3rd, Tran NK, Tzimenatos LS, Michael Dean J, Kuppermann N; TIC-TOC Collaborators of the Pediatric Emergency Care Applied Research Network. Traumatic injury clinical trial evaluating tranexamic acid in children (TIC-TOC): study protocol for a pilot randomized controlled trial. Trials. 2018 Oct 30;19(1):593. doi: 10.1186/s13063-018-2974-z. PMID 30376893
- [Result] Nishijima DK, Gosdin M, Naz H, Tancredi DJ, Hewes HA, Myers SR, Stanley RM, Adelson PD, Burd RS, Finkelstein Y, VanBuren J, Casper TC, Kuppermann N; TIC-TOC Collaborators of the Pediatric Emergency Care Applied Research Network (PECARN). Assessment of primary outcome measures for a clinical trial of pediatric hemorrhagic injuries. Am J Emerg Med. 2021 May;43:210-216. doi: 10.1016/j.ajem.2020.03.001. Epub 2020 Mar 9. PMID 32278572
- [Result] Trappey AF 3rd, Thompson KM, Kuppermann N, Stephenson JT, Nuno MA, Hewes HA, Meyers SR, Stanley RM, Galante JM, Nishijima DK; Traumatic Injury Clinical Trial Evaluating Tranexamic Acid in Children (TIC-TOC) Collaborators of the Pediatric Emergency Care Applied Research Network (PECARN). Development of transfusion guidelines for injured children using a Modified Delphi Consensus Process. J Trauma Acute Care Surg. 2019 Oct;87(4):935-943. doi: 10.1097/TA.0000000000002432. PMID 31299040
- [Result] Powers PE, Shore KK, Perez S, Ritley D, Kuppermann N, Holmes JF, Tzimenatos LS, Shawargga H, Nishijima DK. Public Deliberation as a Novel Method for an Exception From Informed Consent Community Consultation. Acad Emerg Med. 2019 Oct;26(10):1158-1168. doi: 10.1111/acem.13827. Epub 2019 Jul 24. PMID 31271691
- [Derived] Patel PA, Wyrobek JA, Butwick AJ, Pivalizza EG, Hare GMT, Mazer CD, Goobie SM. Update on Applications and Limitations of Perioperative Tranexamic Acid. Anesth Analg. 2022 Sep 1;135(3):460-473. doi: 10.1213/ANE.0000000000006039. Epub 2022 Aug 17. PMID 35977357
- See also: TIC-TOC trial website — https://tictoctrial.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid Dose A | Tranexamic Acid Dose B | Placebo
Started | 9 | 10 | 12
Completed | 9 | 10 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid Dose A | Tranexamic Acid Dose B | Placebo | Total
Number analyzed (Participants) | 9 | 10 | 12 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.6 (4.4) | 10.7 (4.0) | 9.2 (6.1) | 10.7 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 9
  Male | 5 | 8 | 9 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 4 | 8
  White | 4 | 6 | 6 | 16
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 2 | 2 | 1 | 5
Injury Type [Count of Participants; unit: Participants]
  TBI | 4 | 5 | 7 | 16
  Torso | 5 | 5 | 5 | 15
Method of transport to the emergency department [Count of Participants; unit: Participants]
  EMS air | 1 | 4 | 5 | 10
  EMS ground | 8 | 5 | 4 | 17
  Private vehicle/walk-in | 0 | 0 | 1 | 1
  Interfacility transfer | 0 | 0 | 1 | 1
  Multiple methods of transportation | 0 | 1 | 1 | 2
Time from injury to emergency department arrival [Mean (Standard Deviation); unit: hours] | 0.8 (0.5) | 1.2 (0.5) | 1.1 (0.8) | 1.0 (0.6)
Time from injury to randomization [Mean (Standard Deviation); unit: hours] | 2.3 (0.5) | 2.5 (0.4) | 2.4 (0.7) | 2.4 (0.6)
Primary mechanism of injury [Count of Participants; unit: Participants]
  Fall from greater than standing height | 1 | 2 | 2 | 5
  MVC | 3 | 4 | 2 | 9
  Pedestrian/bicyclist hit by moving vehicle | 1 | 0 | 3 | 4
  Gun-shot wound | 2 | 0 | 2 | 4
  Recreational vehicle injury | 0 | 1 | 0 | 1
  Sport-related injury | 2 | 1 | 2 | 5
  Other | 0 | 2 | 1 | 3
Initial Glasgow Coma Scale score (3 to 15) [Median (Inter-Quartile Range); unit: units on a scale] — Scale is 3 to 15; lower scores represent more severe traumatic brain injury
  units on a scale
    TBI/Both | 13 [10 to 13] | 11 [7 to 13] | 3 [3 to 13] | 9 [3 to 13]
    Torso | 15 [14 to 15] | 15 [14 to 15] | 15 [9 to 15] | 15 [9 to 15]
Emergency department disposition [Count of Participants; unit: Participants]
  Operating room | 3 | 1 | 3 | 7
  Admit | 6 | 9 | 9 | 24
Patient received craniotomy or craniectomy [Count of Participants; unit: Participants] | 0 | 1 | 2 | 3
Patient received an intracranial pressure monitor [Count of Participants; unit: Participants] | 0 | 1 | 3 | 4
Patient received a laparotomy [Count of Participants; unit: Participants] | 3 | 2 | 3 | 8
Patient received a thoracotomy [Count of Participants; unit: Participants] | 1 | 0 | 1 | 2
Length of hospitalization [Mean (Standard Deviation); unit: days] | 8.3 (8.0) | 13.6 (14.7) | 22.3 (28.2) | 15.4 (20.2)
Injury Severity Scale score (0 to 75) [Mean (Standard Deviation); unit: units on a scale] — Scale is 0 to 75 with higher scores representing more severe injury
  units on a scale | 15.1 (5.8) | 15.2 (5.7) | 13.8 (5.7) | 14.6 (5.6)
Presence of peritoneal free fluid on initial focused assessment with sonography for trauma exam [Count of Participants; unit: Participants] | 1 | 2 | 1 | 4
pH [Mean (Standard Deviation); unit: units on a scale] | 7.3 (0.1) | 7.3 (0.1) | 7.3 (0.1) | 7.3 (0.1)
Serum bicarbonate [Mean (Standard Deviation); unit: mmol/L] | 20.4 (2.2) | 22.0 (1.7) | 21.5 (3.2) | 21.4 (2.5)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.7 (0.2) | 0.6 (0.2) | 0.6 (0.3) | 0.7 (0.3)
International Normalized Ratio [Mean (Standard Deviation); unit: ratio] — Normal range is 0.8 to 1.1
  ratio | 1.1 (0.1) | 1.1 (0.2) | 1.2 (0.2) | 1.1 (0.2)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 13.0 (1.1) | 13.1 (1.9) | 12.5 (2.0) | 12.8 (1.7)
Platelets [Mean (Standard Deviation); unit: platelets per microliter] | 323.5 (117.9) | 285.0 (136.5) | 374.7 (138.7) | 329.7 (133.6)
Glomerular filtration rate () [Count of Participants; unit: Participants]
  Moderate renal dysfunction | 0 | 0 | 1 | 1
  Normal renal function | 9 | 10 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Quality of Life Inventory (PedsQL)
Description: Neurocognitive functioning and quality-of-life measures; range from 0 to 100 quality of life units with higher scores representing better outcomes. Measurements occur at 1 week, 1 month, 3 months, and 6 months to generate an area under the curve of quality of life units.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Quality of life units * months
Arm/Group | Tranexamic Acid Dose A | Tranexamic Acid Dose B | Placebo
Number analyzed (Participants) | 9 | 10 | 12
Quality of life units * months | 64.9 (19.0) | 60.2 (12.3) | 67.2 (20.0)

2. Primary Outcome: Pediatric Quality of Life Inventory (PedsQL)
Description: Neurocognitive functioning and quality-of-life measures; range from 0 to 100 with higher scores representing better outcomes
Time Frame: 1 week, 1 month, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tranexamic Acid Dose A | Tranexamic Acid Dose B | Placebo
Number analyzed (Participants) | 9 | 10 | 12
units on a scale
  1 week | 43.7 (24.0) | 52.4 (20.1) | 57.9 (28.6)
  1 month | 57.0 (19.8) | 61.5 (16.9) | 60.5 (27.9)
  3 months | 77.3 (23.6) | 77.5 (18.5) | 68.9 (22.5)
  6 months | 81.6 (23.0) | 84.3 (9.9) | 68.9 (25.9)

3. Secondary Outcome: Glasgow Outcome Scale-Extended (GOS-E) Peds
Description: Global functioning; range is 1 to 8 with higher scores representing better outcomes; 1=death, 2=vegetative state, 3=lower severe disability, 4=upper severe disability, 5=lower moderate disability, 6=upper moderate disability, 7=lower good recovery, 8=upper good recovery
Time Frame: 1 week, 1 month, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tranexamic Acid Dose A | Tranexamic Acid Dose B | Placebo
Number analyzed (Participants) | 9 | 10 | 12
score on a scale
  1 week | 4.6 (2.3) | 5.2 (1.8) | 5.3 (2.2)
  1 month | 4.9 (2.0) | 5.1 (1.4) | 4.5 (2.2)
  3 months | 3.8 (2.3) | 4.6 (1.3) | 4.2 (2.4)
  6 months | 3.7 (2.6) | 2.9 (2.3) | 4.3 (2.3)

4. Secondary Outcome: Digit Span Recall Test
Description: Test of working memory; higher scores represent a better outcome, range from 0 to infinity
Time Frame: 1 week, 1 month, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tranexamic Acid Dose A | Tranexamic Acid Dose B | Placebo
Number analyzed (Participants) | 9 | 10 | 12
score on a scale
  Total forward digit span, 1 week | 8.4 (1.7) | 8.4 (4.3) | 8.8 (2.8)
  Total backward digit span, 1 week | 6.0 (1.6) | 6.0 (3.3) | 7.3 (1.0)
  Total forward digit span, 1 month | 7.2 (1.9) | 7.9 (3.7) | 7.5 (2.6)
  Total backward digit span, 1 month | 6.2 (1.8) | 6.2 (1.3) | 5.3 (2.6)
  Total forward digit span, 3 months | 9.1 (3.6) | 10.4 (1.5) | 8.6 (2.5)
  Total backward digit span, 3 months | 8.7 (3.6) | 7.8 (0.8) | 6.5 (1.1)
  Total forward digit span, 6 months | 11.7 (3.9) | 10.0 (2.4) | 8.4 (2.3)
  Total backward digit span, 6 months | 10.4 (4.1) | 6.0 (2.4) | 5.8 (2.9)

5. Secondary Outcome: Blood Transfusion
Description: Total volume of packed red blood cells, platelets, fresh frozen plasma, and cryoprecipitate
Time Frame: First 48 hours after randomization
Population: Torso and Both groups
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Tranexamic Acid Dose A | Tranexamic Acid Dose B | Placebo
Number analyzed (Participants) | 5 | 5 | 5
ml | 367.4 (821.5) | 150.4 (214.1) | 303.6 (571.9)

6. Secondary Outcome: Intracranial Hemorrhage Progression
Description: Intracranial hemorrhage progression on cranial computed tomography (CT) imaging; hemorrhage will be measured using the ABC/2 volume estimation and relative to the total brain volume (calculated by the XYZ/2 volume estimation); more intracranial hemorrhage progression represents a worse outcome. Change is calculated as the difference between the baseline and repeat cranial CT imaging. The repeat CT is conducted 24 hours (±6 hours) after the baseline CT.
Time Frame: 24 hours (±6 hours)
Population: Brain Injury and Both groups
Measure: Mean (Standard Deviation); unit: Proportional change
Arm/Group | Tranexamic Acid Dose A | Tranexamic Acid Dose B | Placebo
Number analyzed (Participants) | 4 | 4 | 7
Proportional change | 0.003 (0.004) | 0.001 (0.001) | 0.003 (0.013)

7. Secondary Outcome: Number of Participants With Any Non-cerebral Venous or Arterial Thrombosis
Description: Any non-cerebral venous or arterial thrombosis on standard diagnostic imaging post-randomization
Time Frame: Day 7 of hospitalization or hospital discharge (whichever comes first)
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Dose A | Tranexamic Acid Dose B | Placebo
Number analyzed (Participants) | 9 | 10 | 12
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Seizures
Description: Clinical or electroencephalogram-documented
Time Frame: 24 hours after receiving drug
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Dose A | Tranexamic Acid Dose B | Placebo
Number analyzed (Participants) | 9 | 10 | 12
Participants | 0 | 0 | 1

9. Secondary Outcome: Biomarker Testing
Description: Changes in coagulation biomarkers due to study intervention
Time Frame: Baseline and completion of 8 hour infusion
Population: Data were not collected
Arm/Group | Tranexamic Acid Dose A | Tranexamic Acid Dose B | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event; defined as any untoward medical occurrence experienced by a subject; may constitute a disease, a set of related signs or symptoms, or a single sign or symptom
Arm/Group | Tranexamic Acid Dose A | Tranexamic Acid Dose B | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 1/12
Other Adverse Events (participants affected / at risk) | 9/9 | 10/10 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid Dose A (N=9) | Tranexamic Acid Dose B (N=10) | Placebo (N=12)
Seizure (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid Dose A (N=9) | Tranexamic Acid Dose B (N=10) | Placebo (N=12)
Adverse Event (General disorders) | 9 | 10 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT02840097/Prot_SAP_001.pdf